CLINICAL TRIAL: NCT02695459
Title: Phase II Study of Cisplatinum and Everolimus in Patients With Metastatic or Unresectable Neuroendocrine Carcinomas (NEC) of Extrapulmonary Origin
Brief Title: Cisplatinum and Everolimus in Patients With Metastatic or Unresectable NEC of Extrapulmonary Origin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14NEC
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Neuroendocrine Carcinomas
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Cisplatin; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cisplatinum and everolimus (Experimental): Cisplatinum : 75 mg/m2 days 1,iv Everolimus : 7.5 mg daily: days 1-21 orally
  Interventions: Drug: cisplatinum and everolimus

INTERVENTIONS:
Drug: cisplatinum and everolimus — Cisplatinum : 75 mg/m2 days 1,iv Everolimus : 7.5 mg daily: days 1-21 orally
  Other Names: cisplatinum; everolimus

SUMMARY:
Phase II, open-label, multicentre national study. Patients with metastatic neuroendocrine carcinomas of extrapulmonary origin will be eligible. Treatment will be performed as indicated in the section "Investigational drug and reference therapy". Cisplatinum and everolimus dosing is based upon earlier phase 1 studies (Fury et al. 2012). CTs will be done at 9 weekly intervals (after 3 courses of chemotherapy;). Patients will be treated until documented progression according to RECIST 1.1. Enrolment is expected to take between 14 - 16 months. The total study duration is estimated to be 2 to 3 years until publication. Three NET centres in The Netherlands will participate, (Erasmus Medical Center in Rotterdam, Netherlands Cancer Institute in Amsterdam and , the University Medical Center of Groningen) A pre-treatment (and optional post-treatment) tumour biopsy will be included for DNA/RNA analyses and organoid culture. An additional 5cc of blood will be withdrawn as a germline DNA reference. A second 5 cc of blood will be included for measuring circulating tumour transcripts to identify all types of GEP-NET (NETTest).

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed unresectable locally advanced and/or metastatic NEC of extrapulmonary origin (WHO 2010 classification; Ki67 >20 %) where no curative (chemoradiation) treatment options are available(including merkel cell carcinoma).
2. Measurable disease according to RECIST 1.1, on CT-scan or MRI
3. ECOG Performance status 0-2 (see Appendix 2)
4. Adequate bone marrow function as shown by: ANC≥1.5 x 109/L, Platelets ≥100 x 109/L, Hb >6 mmol/L
5. Adequate liver function as shown by:

   * Total serum bilirubin ≤1.5 ULN
   * ALT and AST ≤2.5x ULN (≤5x ULN in patients with liver metastases)
6. Adequate renal function: calculated creatinin clearance > 60ml/min. (Cockcroft-Gault formula)
7. Life expectancy of at least 3 months.
8. Male or female age ≥ 18 years.
9. Signed informed consent.
10. Able to swallow and retain oral medication.
11. Locally advanced or metastatic lesion(s) of which a histological biopsy can safely be obtained:

    * Patients with safely accessible locally advanced or metastatic lesion(s) including bone lesions.
    * Patients not known with bleeding disorders (such as hemophilia) or bleeding complications from biopsies, dental procedures or surgeries.
    * Patients not using any anti-coagulant medication at the time of biopsy: all aspirin derivatives, NSAID's, coumarines, platelet function inhibitors, heparins (including LMWHs) and oral factor Xa inhibitors are not allowed, unless medication can either be safely stopped or counteracted.
    * Adequate coagulation status as measured by:

      * PT < 1.5 x ULN or PT-INR < 1.5
      * APTT < 1.5 x ULN
      * On the day of biopsy in patients using coumarines: PT-INR < 1.5
12. Patients not known with contraindications for lidocaine (or its derivatives)

Exclusion Criteria:

1. Previous chemotherapy for metastatic or unresectable NEC of extrapulmonary origin. (prior peri-operative chemotherapy or chemoradiation for curative intention is allowed if at least 6 months have elapsed between completion of this therapy and enrolment into the study).
2. Prior therapy with mTOR inhibitors (e.g. sirolimus, temsirolimus, deforolimus, everolimus)
3. Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.
4. Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus) or cisplatinum
5. Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
6. Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
7. Patients who have any severe and/or uncontrolled medical conditions such as: a. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to randomization, serious uncontrolled cardiac arrhythmia and poorly controlled hypertension (systolic BP >180 mmHg or diastolic BP >100 mmHg);. b. active or uncontrolled severe infection, c. liver disease such as cirrhosis, decompensated liver disease, and known history chronic hepatitis d. known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air), e. active, bleeding diathesis;
8. Chronic treatment with corticosteroids or other immunosuppressive agents
9. Known history of HIV seropositivity
10. Pregnant or nursing (lactating) women
11. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 6 months after stopping study treatment.
12. Sexually active males, unless they use a condom during intercourse while taking study medication and for 6 months after stopping study medication.
13. Patients with dyspnoea at rest due to complications of advanced malignancy or other disease, or who require supportive oxygen therapy.
14. History or clinical evidence of brain metastases.
15. Any investigational drug treatment within 4 weeks of start of study treatment.
16. Radiotherapy within 4 weeks of start of study treatment (2 week interval allowed if palliative radiotherapy given to bone metastatic site peripherally and patient recovered from any acute toxicity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
disease control rate | every 9 weeks until up to 16 months
  patients having a complete response, partial response or stable disease are considered successes

SECONDARY OUTCOMES:
time to relapse | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
overall survival | Time from registration until the date of death from any cause, assessed up to 60 months
Effect on the markers chromogranin A (CgA) and neuron-specific enolase (NSE); | from registration in the study markers will be taken every cycle until a maximum of 6 cycles is reached (cycle is every 3 weeks), until a maximum of 18 weeks.
Safety of everolimus in combination with cisplatin (AEs according to CTCAE v4.0) | up to 30 days after end of treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
discovery of biomarkers (including circulating neuroendocrine tumour transcripts: NETTest) for treatment response; | during the 6 cycles of treatment until 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: M. Tesselaar, MD, Principal Investigator — NKI-AvL
Locations (3):
- Netherlands (3):
  - NKI-AVL, Amsterdam
  - UMCG, Groningen
  - Erasmus Medisch Centrum, Rotterdam

REFERENCES:
- [Derived] Levy S, Verbeek WHM, Eskens FALM, van den Berg JG, de Groot DJA, van Leerdam ME, Tesselaar MET. First-line everolimus and cisplatin in patients with advanced extrapulmonary neuroendocrine carcinoma: a nationwide phase 2 single-arm clinical trial. Ther Adv Med Oncol. 2022 Feb 27;14:17588359221077088. doi: 10.1177/17588359221077088. eCollection 2022. PMID 35251315